CLINICAL TRIAL: NCT02483910
Title: Efficacy of the Direct Instruction Language for Learning Program to Promote Expressive and Receptive Language in Children With Autism Spectrum Disorder
Brief Title: Direct Instruction Language for Learning in Autism Spectrum Disorder
Acronym: DILLASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lawrence Scahill, MSN, PhD, Professor of Pediatrics, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00081144; AR140208 (Other: CDMRP)
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder; Moderate Language Delay
Keywords: School-age children; Pediatrics; Direct Instruction-Language for Learning
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DI-LL via telehealth (Experimental): Subjects with autism spectrum disorder (ASD) plus moderate language between 4 years and 7 years 11 months will be randomly assigned to receive Direct Instruction-Language for Learning (DI-LL) for 40-48 sessions (roughly twice a week for 24 weeks). Subjects in this arm will be allowed to continue ongoing treatment during the randomized phase of the study
  Interventions: Behavioral: Direct Instruction-Language for Learning (DI-LL) via telehealth (e.g., Zoom or WebEx); Behavioral: Standard of care delivered via telehealth (e.g., Zoom or WebEx)
- Standard of care delivered via telehealth (Active Comparator): Subjects with (ASD) plus moderate language between 4 years and 7 years 11 months will be randomly assigned to continue treatment as usual (TAU) for 24 weeks.
  NOTE: after the randomized trial, subjects who do not show a positive response at Week 24, will be offered Direct Instruction-Language for Learning (DI-LL) for 24 weeks.
  Interventions: Behavioral: Standard of care delivered via telehealth (e.g., Zoom or WebEx)

INTERVENTIONS:
Behavioral: Direct Instruction-Language for Learning (DI-LL) via telehealth (e.g., Zoom or WebEx) — DI-LL is composed of up to 150 lessons (15 sets of 10 lessons each - e.g., lessons 1-10, 11-20, 21-30, etc.) that build on one another. The program uses demonstrations and pictures to expand vocabulary and teach language skills to children in manageable steps. The curriculum focuses on teaching spoken language across six areas: actions, description of objects, general information, standardized prompts ("show me" or "point to" or "say the whole thing"), classification, and problem-solving strategies. For example, DI-LL moves from the identification of familiar objects to the description and classification of these objects. Children learn the precise meaning of both familiar and new concepts and use these concepts in statements and questions. The DI-LL also incorporates 15 assessment tests (one for each set of 10 lessons). These assessment tests are given after each set of 10 lessons to confirm mastery of the material and the child's readiness to move on to the next set of 10 lessons.
  Other Names: Due to the shut down imposed by the coronavirus delivery of the intervention is via telehealth (e.g., Zoom or WebEx)
  Arms: DI-LL via telehealth
Behavioral: Standard of care delivered via telehealth (e.g., Zoom or WebEx) — Usual care including speech therapy in school, community or both
  Other Names: Due to the shut down imposed by the coronavirus delivery of the intervention is via telehealth (e.g., Zoom or WebEx)

SUMMARY:
The purpose of this study is to test whether Direct Instruction - Language for Learning (DI-LL) is an effective way to teach language skills to children with autism spectrum disorder (ASD) and moderate language delay. Direct Instruction - Language for Learning (DI-LL) uses face to face instruction and specific lessons to teach children language skills. This method has been used previously in children with language delays, but it has not been carefully studied in children with autism spectrum disorder. This study will compare DI-LL and ongoing treatment as usual to treatment as usual (speech therapy, language services, etc.) alone.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a chronic condition of early childhood onset defined by social impairment and repetitive behavior, and affecting 6 to 14 children per 1000 worldwide. Language and communication impairments are among the most common parental concerns about their children with ASD. Untreated language impairments are also predictive of negative long-term outcomes for children with ASD. Direct Instruction-Language for Learning (DI-LL) is a commercially available intervention package that has demonstrated effectiveness in children with language delays due to disadvantaged backgrounds, learning disabilities, or a primary language disorder - but it has not been carefully studied in ASD. This study will test the efficacy of DI-LL in young school-age children with ASD and moderate language delay. DI-LL is a structured, relatively inexpensive intervention designed to promote a range of language skills. It offers a comprehensive, carefully sequenced, brisk-paced program designed to teach a range of language skills to children with language impairments. A key strength of DI-LL is that it can be implemented by educators, psychologists, speech pathologists, behavior therapists without requiring deep expertise in behavioral interventions for ASD.

100 participants, ages 4 to 7 years, 11 months, will be randomly assigned to either DI-LL or Treatment as Usual (TAU). Children randomly assigned to DI-LL will be allowed to continue in ongoing treatments as well. Forty to 42 treatment sessions will occur across 24 weeks with post-treatment follow up visits at Weeks 36 and 48 for subjects in DI-LL. Negative responders to TAU at Week 24 will be offered treatment with DI-LL for 24 weeks. This study is designed to compare DI-LL and TAU on two standardized tests of language function; overall improvement rated by a blinded clinician; and the number of spoken words in a structured laboratory setting via direct observation - again blind to treatment assignment. The intent to treat approach will be used in efficacy analysis and adverse events will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following age and Clinical Evaluation of Language Fundamentals -version 4 (CELF-4) or Clinical Evaluation of Language Fundamentals Preschool-2 (CELF-P) score combinations:

  * Males and females > 4 years and < 7 years 11 months of age in with a score < 80 on the CELF-4 or the CELF-P, or
  * Males and females > 5 years and < 7 years 11 months of age with a score > 40 on the CELF-4, or
  * Males and females > 4 years and < 6 years 5 months of age with a score > 45 CELF-P
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of autism spectrum disorder (ASD) established by clinical assessment, corroborated by the Social Communication Questionnaire and the Autism Diagnostic Observational Schedule
* A score < 80 on the Core Language score of the Clinical Evaluation of Language Fundamentals - 4 if > 6 years 5 months
* Stable educational plan with no planned changes in the intensity of treatment for 6 months
* Stable community treatment program (e.g., speech therapy or occupational therapy) with no planned changes in the treatment for 6 months. (Otherwise eligible subjects with anticipated changes in their community treatment program in the near term will be invited to return when the transition has been accomplished).
* English is spoken in the home and at least one parent is able to read, write and speak English
* Psychotropic medication free or on stable psychotropic medication (no changes in past 6 weeks and no planned changes for the next 6 months)

Exclusion Criteria:

* Presence of a known serious medical condition in the child (based on medical history) that would interfere with child ability to participate in the study
* On examination, child has less than 5 words and unable to imitate at least 5 words
* Children > 6 years 5 months who achieve a score of 40 on the CELF-4 (and judged to be below 40 by the speech language pathologist)
* Presence of a current serious behavioral problem or psychiatric condition in the child that would require another treatment (e.g., psychotic disorder, major depression, moderate or greater aggression, severe disruptive behavior) based on all available information collected at screening
* Currently receiving Direct Instruction Language for Learning (DI-LL) or participation in a DI-LL program in the past 2 years
* Primary mode of communication is a speech generating device (e.g., DynaVox, Gotalk, Proloquo2go)
* On psychotropic medication, but regimen is not stable (Once stabilized, eligibility could be reconsidered.)

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical Evaluation of Language Fundamentals-4 (CELF-4) Score | Baseline, Week 24, Week 48
  The CELF-4 English Version will be administered to assess the participant's (aged 5-8 years) receptive and expressive language skills.The Core Language score quantifies a participant's overall language performance. The standard score for the Core Language scale is based on a mean of 100 with a standard deviation of 15 (average range of 85-115). The higher the score, the better the language function of the participant.
Change in Clinical Evaluation of Language Fundamentals-Preschool 2 (CELF-P) Score | Baseline, Week 24, Week 48
  The CELF-P English Version will be administered to assess the preschool-aged participant's receptive and expressive language skills.The Core Language score quantifies a participant's overall language performance. The standard score for the Core Language scale is based on a mean of 100 with a standard deviation of 15 (average range of 85-115). The higher the score, the better the language function of the participant.

SECONDARY OUTCOMES:
Improvement item of the Clinical Global Impression scale (CGI-I) | Baseline, Week 24, Week 48
  An independent evaluator, who is blind to treatment assignment, will rate the CGI-I using all available information (e.g. Parent Nominated Problems and parent ratings) to assess overall improvement from baseline. It involves a seven-point scale, from 1 "very much improved" through 4 "no change" and 7 "very much worse." By convention, scores of Much Improved (score of 2) or Very Much Improved (score of 1) are used to define positive response; all other scores result in a classification of negative response.

OTHER OUTCOMES:
Change in Growth Scale Value score of the Expressive Vocabulary Test-2 (EVT-2) | Baseline, Week 24
  The EVT-2 will be administered to measure expressive vocabulary and word retrieval for Standard American English. The Growth Scale Value (GSV) is used to monitor growth on the EVT. The GSV is a score that tracks vocabulary over time. An increase in vocabulary will result in a higher GSV score.
Change in Parent-rated Vineland Adaptive Behavior Scales II (Vineland-II) | Baseline, Week 24, Week 48
  Vineland-II is a measure of adaptive skills in every day life. Scores may range from 20-160 with an average of 100 with a standard deviation of 15. Higher scores indicate better adaptive functioning.
Change in Parenting Stress Index - Short Form (PSI-SF) | Baseline, Week 24
  The PSI-SF is a parent-report questionnaire of parental stress, parent-child interaction style, and difficult child behaviour that will be used to measure changes in parental stress. It is a 36-item questionnaire for families of children 12 years of age and younger. Each of these items is scored using the following 5-point scale: 1 (strongly agree) to 5 (strongly disagree). The total stress score is a composite of the three subscales. Higher scores indicate higher parental stress.
Change in Caregiver Strain Questionnaire (CGSC) | Baseline, Week 24
  The CGSC measures the impact of having a child with ASD on the family. The questionnaire includes 21 items that assess three dimensions of caregiver strain: objective strain, internalized subjective strain, and externalized subjective strain. Each item is rated on a 5-point scale ranging from 1(not at all a problem) to 5 (very much a problem). The total score can range from a minimum of 0 - no strain at all, to 110 all items rated as very much.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, MSN, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center - Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scahill L, Shillingsburg MA, Ousley O, Pileggi ML, Kilbourne RL, Buckley D, Gillespie SE, McCracken C. A Randomized Trial of Direct Instruction Language for Learning in Children With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2022 Jun;61(6):772-781. doi: 10.1016/j.jaac.2021.11.034. Epub 2022 Jan 31. PMID 35093490

DOCUMENTS (1):
  • Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT02483910/ICF_000.pdf